CLINICAL TRIAL: NCT00160329
Title: The De-Escalate Trial: Atazanavir or Atazanavir/Ritonavir Substitution for Ritonavir Boosted PI Therapy in HIV-Infected Individuals Experiencing Ongoing HIV Viremia and Hyperlipidemia: A Randomized Controlled Pilot Study
Brief Title: Atazanavir or Boosted Atazanavir Substitution for Ritonavir Boosted PI in Patients With Hyperlipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Andrew Zolopa, Stanford university
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: De-Escalate Trial; IRB # 79603 (Other: Stanford University); Spo# 29750 (Other: Stanford University)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Hyperlipidemia; HIV Infections
MeSH Terms: conditions — Hyperlipidemias; HIV Infections | interventions — Atazanavir Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Atazanavir — 300 mg with ritonavir boosting or 400 mg without
  Other Names: Reyataz

SUMMARY:
The study is looking to compare the impact of lipid levels and HIV viral loads between three different drug regimens: Continuing current regimen (ritonavir boosted regimen), Switching to Atazanavir, or Switching to Atazanavir in combination to Ritonavir.

DETAILED DESCRIPTION:
Study Overview

This is a randomized controlled pilot study to compare the safety and efficacy of substitution of atazanavir (ATV) or ATV/RTV for ritonavir boosted PI in patients with ongoing viremia who are experiencing hyperlipidemia and/or requiring treatment with lipid lowering agents. In this study 60 subjects on a ritonavir boosted PI-containing antiretroviral regimen who are experiencing hyperlipidemia and ongoing HIV viremia will be randomized in a 1:1:1 ratio to either switch the ritonavir boosted PI component of the antiretroviral regimen to ATV or ATV/RTV, or continue the ritonavir boosted PI-based regimen.

No other changes in the antiretroviral regimen will be allowed for the first 12 weeks. Thereafter, the investigator may change background ARVs based on the results of the screening resistance test. No new class of antiretrovirals will be allowed to be added through 48 weeks. Subjects will be monitored closely over 48 weeks with careful assessment of CD4 profile, viral loads and lipid profiles as well as drug resistance and replication capacity. Stopping rules will be implemented based on CD4 and viral load profile to ensure subject safety. The objective of this study is to determine whether protease inhibitor regimens that have less of an adverse impact on lipid profiles can maintain a stable CD4 profile compared to standard ritonavir boosted PI regimens.

Background

Antiretroviral regimens that include ritonavir-boosted protease inhibitors are commonly recommended and prescribed, particularly in patients with some degree of drug resistance. Despite the potency of boosted regimens, many HIV-infected patients receiving these regimens have incomplete viral suppression and yet maintain clinical stability and CD4 counts above nadir levels: the so called 'CD4/HIV disconnect' state. It is likely that this state of CD4/HIV discordance is due in part to the maintenance of drug resistant HIV virus that is relatively unfit, that is its replication capacity and ability to infect and destroy CD4 cells is compromised. The selective pressure exerted by antiretroviral therapy appears to be important in maintaining these drug resistant but relatively unfit quasispecies. It has been shown that even patients with CD4 counts below 50 cells/cc and ongoing viremia maintain a clinical benefit from continued therapy.

Unfortunately, lipid abnormalities are commonly seen in patients receiving boosted PI regimens. For example, in a clinical trial in which lopinavir/ritonavir (LPV/r) was given to treatment naïve subjects, approximately 1/3 developed grade 2 or higher lipid abnormalities over 48 weeks. There is a growing concern that these lipid abnormalities will increase the risk of cardiovascular morbidity and mortality. In fact, recent data suggest an increased risk of cardiovascular morbidity and mortality related to HIV infection and/or antiretroviral therapy. There are increasing efforts directed at minimizing long-term toxicities of antiretroviral therapy while maintaining its clinical benefit. (Witness the high degree of interest in treatment interruptions as a strategy to limit toxicities associated with long-term antiretroviral therapy.)

Atazanavir (ATV), a recently approved PI, appears to have little to no impact on the lipid profile in subjects enrolled in clinical trials. Other advantages with atazanavir are its dosing schedule and overall tolerability. Furthermore, recent studies using ritonavir-boosted ATV also show favorable lipid effects compared to LPV/r. Ritonavir boosting provides higher drug levels and therefore may improve the potency of ATV, especially against PI-resistant virus.

ELIGIBILITY:
Inclusion Criteria:

Stable primary care

1. Male or Female HIV + adults > 18 years of age.
2. Subjects who are receiving a ritonavir-boosted PI-containing regimen.
3. Subjects who are on a stable antiretroviral regimen for > 3 months.
4. Subjects who have a plasma viral load > 1,000 and < 100,000 c/mL.
5. Protease Inhibitor (PI) resistance: Subjects must have a minimum of 3 of the following PI-mutations (10, 20, 46, 47, 48, 50V, 54, 71, 82, 84, 90).
6. Subjects who have a CD4 > 100 cells/cc.
7. Subjects who are experiencing hyperlipidemia :
8. Total cholesterol > 240 mg/dL, or
9. LDL > 160 mg/dL, or
10. Fasting triglycerides > 200 mg/dL, or
11. On lipid lowering drugs.
12. All women of reproductive potential (who have not reached menopause or undergone hysterectomy, bilateral oophorectomy, or tubal ligation) must have a negative serum or urine ²-HCG pregnancy test performed within 48 hours of entry.

    Female study volunteers who are not of reproductive potential (who have reached menopause or undergone hysterectomy, bilateral oophorectomy, or tubal ligation) or whose male partner has undergone successful vasectomy with documented azoospermia or has documented azoospermia for any other reason, are eligible without requiring the use of contraception. Acceptable documentation of menopause, sterilization, and azoospermia are as follows:
13. Written or oral documentation communicated by clinician or clinician's staff of one of the following:

    1. Physician report/letter
    2. Operative report or other source documentation in the patient record
    3. Discharge summary
    4. Laboratory report of azoospermia (required for acceptable documentation of successful vasectomy)
    5. FSH measurement elevated into the menopausal range as established by the reporting laboratory. Exclusion Criteria:1. Women who are pregnant or breast feeding.

2. Subjects who use substances or with a mental health condition that would in the opinion of the treating clinician interfere with the ability of the subject to comply with study treatment and monitoring.

3. Subjects who have significant liver disease defined as AST (SGOT) and ALT (SGPT) > 5 x ULN.

4. Subjects who have a history of an acute opportunistic infection within 8 weeks prior to study screening. Chronic infections will not be excluded.

5. Subjects who have received a vaccination within 2 weeks prior to study screening.

6. Subjects who are receiving experimental ARV therapy.

7. Subjects who are receiving systemic chemotherapy.

8. Subjects who are receiving IL-2 or IFN-alpha.

9. Subjects who are receiving GM-CSF.

10. Subjects who have any grade 3-4 laboratory abnormality or clinical AE, other than lipid abnormalities.

11. Prior use of Atazanavir

12. Subjects who have a history of

1. Symptomatic heart block
2. 3rd degree heart block, even if asymptomatic
3. Pre-excitation syndromes
4. Heart rate < 40 bpm
5. Ventricular pause length > 3 sec
6. QTc > 500 msec
7. History of syncope of undetermined origin
8. Cardiomyopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-01; Primary Completion 2007-04 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Compare the three arms (ATV, ATV/r and continued ritonavir boosted-PI) in the following primary endpoint: % subjects who have normal serum lipid profile off lipid lowering agents and maintain CD4 counts > 75% of baseline line values. | 48 weeks

SECONDARY OUTCOMES:
% subjects with serum lipids within normal limits at week 48 off of any lipid lowering agent. | 48 weeks
% subjects who maintain CD4 counts > 75% of baseline values at week 48. | 48 weeks
Compare the change in CD4 count and CD4 % at 24 and 48 weeks between the three study arms.1.2.4Compare HIV plasma viral load profile over 24 and 48 weeks as DAVG between the three study arms. | 24 and 48 weeks
Compare lipid profile over 48 weeks, change in total cholesterol, TC/HDL ratio and triglycerides. | 48 weeks
Compare the evolution of genotypic and phenotypic drug resistance over 12 and 48 weeks between the three arms. | 12 and 48 weeks
Compare the evolution of viral fitness as measured by replication capacity assay at 12 and 48 weeks between the three arms. | 12 and 48 weeks
Explore determinates of viral fitness and the relationship of viral fitness with the 'CD4/VL disconnect' state. | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andrew R Zolopa, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States